CLINICAL TRIAL: NCT07372443
Title: Usefulness of Photobio-modulation in the Prevention and Management of Oral Mucositis in Pediatric Patients Undergoing Antineoplastic Treatment: Randomized Clinical Trial
Brief Title: Photobiomodulation in the Prevention and Management of Oral Mucositis in Children
Acronym: PBMOM-PEDMX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Guanajuato (Other)
Responsible Party: Principal Investigator, Mariana Paulina Rodríguez Vargas, Principal Investigator, Universidad de Guanajuato
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MX-UG-PBM-PED-2025-001
Record Dates: First submitted 2026-01-09; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Oral Mucositis; Chemotherapy Effect; Pediatric Cancer
Keywords: Photobiomodulation
MeSH Terms: conditions — Stomatitis; Neoplasms | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Simple-blind randomized clinical trial. Two arms: Treatment (parallel design). Prevention (crossover design).
Who Masked: Outcomes Assessor
Masking Description: Blinding: open for the principal investigator, who will be aware of the intervention, and blinded to the evaluator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prevention arm (Experimental): Cross-over design: patients receive both interventions (photobiomodulation in the first phase and are reassigned to receive bioadhesive gel in the second phase), i.e., in successive cycles of chemotherapy, within the first three days of the start of chemotherapy, in the absence of oral mucositis.
  Interventions: Device: Photobiomodulation; Drug: bioadhesive gel
- Treatment (Experimental): Treatment arm: randomization into two groups: one receives photobiomodulation, and the other receives bioadhesive gel, in the presence of oral mucositis.
  Interventions: Device: Photobiomodulation; Drug: bioadhesive gel

INTERVENTIONS:
Device: Photobiomodulation — For the prevention arm, photobiomodulation will be applied three alternate days per week starting on the first three days of chemotherapy. It will be applied to areas such as the corners of the mouth, the lip mucosa, the buccal mucosa, the lateral edges of the tongue, the ventral tongue, the anterior floor of the mouth, and the soft palate. For the treatment arm, photobiomodulation will be applied every other day of the week from the detection of oral mucositis until resolution. The application sites will be the affected mucosal areas, whether they present erythema or ulcerations.
Drug: bioadhesive gel — Application of bioadherent gel Rinse with bioadherent gel, 5 consecutive days, 30 to 60 minutes before each meal. Or apply with a swab in young children who are unable to rinse.

SUMMARY:
Oral mucositis (OM) is a frequent, debilitating complication in pediatric oncology that impairs quality of life, nutrition, hydration, and treatment adherence. This randomized, prospective, single blind trial in Mexico will evaluate photobiomodulation (PBM) versus a conventional bioadhesive gel for prevention and treatment of antineoplastic therapy-induced OM in children aged 4-17 with leukemia, lymphoma, or head and neck tumors. A total of 49 participants will be enrolled. The study has two components: (1) Treatment - parallel comparison of PBM versus bioadhesive gel for established OM; (2) Prevention - crossover design in which patients receive both interventions across successive chemotherapy cycles. PBM will be delivered with a 660 nm device, 40 mW, 10 J/cm². The primary outcome is OM grade by the WHO scale assessed on days 7, 11, 14, and 21. Expected results include reduced OM incidence, severity, duration, and pain with favorable safety and tolerability, supporting standardized PBM protocols in pediatric oncology in Mexico.

DETAILED DESCRIPTION:
Oral mucositis is a common and debilitating adverse effect in pediatric patients undergoing cancer treatment. It significantly affects quality of life, nutrition, hydration, and treatment adherence. Photobiomodulation is a promising non-invasive therapy, but there is limited evidence in the pediatric population, particularly in Mexico. Objective: To evaluate the clinical utility of FBM in the prevention and treatment of OM induced by antineoplastic therapy in pediatric cancer patients, compared to conventional treatment with bioadhesive gel. This is a randomized, single-blind clinical trial in patients aged 4 to 17 years. The design includes two arms: 1) Treatment (parallel design: FBM vs. gel for established OM) and 2) Prevention (crossover design: patients receive both interventions in successive cycles of chemotherapy). The primary outcome will be the degree of OM according to the WHO scale. FBM is expected to significantly reduce the incidence, severity, and duration of OM, as well as the intensity of pain. In addition, scientific evidence will be generated on the implementation of FBM in pediatric oncology in Mexico, with the potential to standardize protocols that improve patients' quality of life and optimize the management of oral complications of antineoplastic treatment.

ELIGIBILITY:
Inclusion Criteria:

Prevention Arm - Inclusion Criteria

* Age 4 to 17 years
* Histopathologic diagnosis of malignant neoplasm: leukemia, lymphoma, or solid tumor of the head and neck.
* Within days 1-3 of the start of any chemotherapy cycle; for leukemia patients, in consolidation phase as defined by protocol.
* No signs of oral mucositis at enrollment.
* Availability and willingness to attend scheduled photobiomodulation (PBM) application sessions.
* Parent/legal guardian signed informed consent and child assent when applicable (≥ 8 years).
* No documented primary immunodeficiency.
* No severe concomitant systemic infection or medical condition that, in the investigator's judgment, contraindicates participation.
* No PBM treatment within 14 days prior to enrollment.
* No history of adverse reactions to light therapies or known photosensitivity.
* No history of seizure disorder or diagnosis of epilepsy.

Treatment Arm - Inclusion Criteria

* Age 4 to 17 years
* Histopathologic diagnosis of malignant neoplasm: leukemia, lymphoma, or solid tumor of the head and neck.
* Currently receiving chemotherapy (any cycle of the regimen).
* Presence of oral mucositis of any grade during chemotherapy, identified within the first 3 days from onset of the mucositis episode.
* Parent/legal guardian signed informed consent and child assent when applicable (≥ 8 years).
* No documented primary immunodeficiency.
* No severe concomitant systemic infection or medical condition that, in the investigator's judgment, contraindicates participation.
* No photobiomodulation (PBM) treatment within 14 days prior to enrollment.
* No history of adverse reactions to light therapies or known photosensitivity.
* No history of seizure disorder or diagnosis of epilepsy.

Exclusion Criteria:

* Documented primary immunodeficiency.
* Severe concomitant systemic infection or unstable medical condition.
* PBM treatment within 14 days prior to enrollment.
* Known photosensitivity or prior adverse reaction to light therapy.
* History of seizures or epilepsy.
* Any condition that, in the investigator's opinion, would interfere with study participation or safety.

Participant Withdrawal Criteria

* Attendance to fewer than 80% of scheduled treatment sessions.
* Any adverse event or persistent discomfort attributed to PBM that leads the participant or guardian to decline further intervention.
* Withdrawal of consent by parent/guardian or assent withdrawal by participant when applicable.
* Development of a new medical condition that, per investigator judgment, contraindicates continuation.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Oral mucositis grade | Days 7, 11, 14, and 21 after intervention initiation for each episode/cycle (each cycle is 14 days)
  Grade of oral mucositis assessed using the World Health Organization (WHO) oral mucositis scale (0-4). Assessments performed by a blinded clinician trained in the scale

SECONDARY OUTCOMES:
Incidence of oral mucositis | Per chemotherapy cycle and overall study period (up to 21 days post intervention).
  Proportion of chemotherapy cycles in which participants develop oral mucositis defined as WHO grade ≥1; assessments by blinded clinician
Oral mucositis Duration outcome | Mesured for each episode during follow-up
  time from onset of WHO grade ≥1 mucositis to resolution to WHO grade 0.

CONTACTS AND LOCATIONS:
Overall Officials: María C Palacios, PhD, Study Director — Universidad de Guanajuato

IPD SHARING:
Plan to Share IPD: No